CLINICAL TRIAL: NCT01698814
Title: A Multicenter, Randomized, Double-Masked, Vehicle-Controlled, Parallel-Group Study Evaluating the Safety of AL-4943A Ophthalmic Solution Administered Once Daily
Brief Title: A Six-Week Safety Study of an Investigational Ophthalmic Solution
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: C-12-028
Record Dates: First submitted 2012-09-27; First posted 2012-10-03 (Estimated); Results first posted 2014-02-28 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-02

CONDITIONS: Allergic Conjunctivitis
Keywords: ocular safety; allergic conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AL-4943A (Experimental): AL-4943A Ophthalmic Solution, one drop instilled in both eyes once daily for up to 6 weeks
  Interventions: Drug: AL-4943A Ophthalmic Solution
- AL-4943A Vehicle (Placebo Comparator): AL-4943A Ophthalmic Solution Vehicle, one drop instilled in both eyes once daily for up to 6 weeks
  Interventions: Drug: AL-4943A Ophthalmic Solution Vehicle

INTERVENTIONS:
Drug: AL-4943A Ophthalmic Solution
  Arms: AL-4943A
Drug: AL-4943A Ophthalmic Solution Vehicle — Inactive ingredients used as placebo
  Arms: AL-4943A Vehicle

SUMMARY:
The purpose of this study was to evaluate the ocular safety of an investigational ophthalmic solution in subjects 2 years of age and older with asymptomatic eyes when administered once daily in both eyes for up to 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to comply with study protocol and follow protocol instructions.
* Adequate birth control methods for the duration of the study.
* Best-corrected visual acuity (BCVA) of 55 or greater in each eye.
* Willing to avoid contact lens wear during each of the study visits; contact lens wear also should be stable and consistent for 1 month prior to Visit 1 and expected to remain the same for the study duration.
* Willing and able to sign an Informed Consent form.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Women of childbearing potential that are pregnant, breastfeeding, or not in agreement to use adequate birth control methods to prevent pregnancy throughout the study.
* Evidence of contact lens care solution related ocular surface damage or giant papillary conjunctivitis (GPC).
* Any ocular infection (bacterial, viral or fungal) or history of ocular Herpes (simplex or zoster) or adenoviral infection in either eye or have had any ocular infection within 30 days prior to Visit 1.
* Using systemic medication(s) on a chronic dosing regimen for less than 30 days or changed dosage of this medication within 30 days prior to Visit 1.
* Current or past history of glaucoma or ocular hypertension.
* History of retinal detachment, diabetic retinopathy, or progressive retinal disease.
* Presence of ocular conditions that may affect the study outcomes.
* Corneal conditions affecting the corneal structure.
* History or evidence of any ocular surgical procedure within 1 year prior to Visit 1.
* Current or recent medical conditions that, in the opinion of the Investigator, would preclude safe participation in the study.
* Prior, current, or anticipated use of ophthalmic agents other than investigational product during study participation.
* Participation in any investigational study within 30 days prior to Visit 1 or concomitantly with this study.
* Known contraindications or hypersensitivities to any of the study medications or their components.
* Other protocol-specified exclusion criteria may apply.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2012-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terri Pasquine, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 15 study centers located in the United States.
Pre-assignment Details: Of the 518 enrolled subjects, 18 subjects were exited from the study as screen failures. This reporting group includes all randomized subjects.
Period: Overall Study
Arm/Group | AL-4943A | AL-4943A Vehicle
Started | 331 | 169
Completed | 329 | 166
Not Completed | 2 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Randomized in error | 1 | 0

BASELINE CHARACTERISTICS:
Population: This reporting group includes all randomized subjects who received study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | AL-4943A | AL-4943A Vehicle | Total
Number analyzed (Participants) | 330 | 169 | 499
Age, Customized [Number; unit: participants]
  2-11 years | 47 | 21 | 68
  12-17 years | 4 | 3 | 7
  18-64 years | 272 | 141 | 413
  ≥65 years | 7 | 4 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 214 | 111 | 325
  Male | 116 | 58 | 174

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: An adverse event was defined as any untoward medical occurrence in a subject administered a study treatment regardless of causal relationship with the treatment. AEs were obtained as solicited comments from the study subjects and as observations by the study Investigator.
Time Frame: An average of 6 weeks
Population: This reporting group includes all randomized subjects who received study medication.
Measure: Number; unit: participants
Arm/Group | AL-4943A | AL-4943A Vehicle
Number analyzed (Participants) | 330 | 169
participants
  Deaths | 0 | 0
  Non-Fatal Serious Adverse Events | 0 | 0
  Discontinuations Due to an Adverse Event | 0 | 2

ADVERSE EVENTS:
Time Frame: Adverse Events (AE) were collected for the duration of the study (3 months). An AE was defined as any untoward medical occurrence in a subject administered a study treatment regardless of causal relationship with the treatment.
Description: This reporting group includes all randomized subjects who received study medication. AEs were obtained as solicited comments from the study subjects and as observations by the study Investigator.
Arm/Group | AL-4943A | AL-4943A Vehicle
Serious Adverse Events (participants affected / at risk) | 0/330 | 0/169
Other Adverse Events (participants affected / at risk) | 0/330 | 0/169

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.